CLINICAL TRIAL: NCT00876031
Title: A Randomised Phase-III Trial of the Cooperative Weichteilsarkom Study Group (CWS) for Localised High-risk Rhabdomyosarcoma and Localised Rhabdomyosarcoma-like Soft Tissue Sarcoma in Children, Adolescents, and Young Adults
Brief Title: Trial for Localised High-risk Rhabdomyosarcoma and Rhabdomyosarcoma-like Soft Tissue Sarcoma
Acronym: CWS-2007-HR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Cooperative Weichteilsarkom Study Group (Other); Deutsche Kinderkrebsstiftung (Other); German Society for Pediatric Oncology and Hematology GPOH gGmbH (Other); Gesellschaft fur Padiatrische Onkologie und Hamatologie - Austria (Other); The Swedish Childhood Solid Tumor Working Group (Unknown); Polish Paediatric Solid Tumours Study Group (Unknown); Swiss Pediatric Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CWS-2007-HR; 4033024 (BfArM) (Other: Bundesinstitut für Arzneimittel und Medizinprodukte); 293/2007AMG1 (Ethikkommission) (Other: Ethics Committee University of Tübingen); 2007-001478-10 (EudraCT Number); A2007/14 (Kinderkrebsstiftung) (Other: German Childhood Cancer Foundation); 498 (Krebsstudienregister) (Registry Identifier: Krebsstudienregister)
Record Dates: First submitted 2009-04-02; First posted 2009-04-06 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Soft Tissue Sarcoma
Keywords: pediatric soft tissue sarcoma; rhabdomyosarcoma; extraosseous Ewing family tumours; synovial sarcoma; undifferentiated sarcoma
MeSH Terms: conditions — Sarcoma; Rhabdomyosarcoma; Sarcoma, Synovial | interventions — trofosfamide; Idarubicin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- O-TIE (Experimental): oral maintenance therapy with trofosfamide, idarubicin, and etoposide
  Interventions: Drug: trofosfamide, idarubicin, etoposide
- control (No Intervention)

INTERVENTIONS:
Drug: trofosfamide, idarubicin, etoposide — oral maintenance therapy for 6 months
  Arms: O-TIE

SUMMARY:
The purpose of this study is to investigate whether the addition of oral maintenance chemotherapy with O-TIE (Etoposide, Idarubicin, Trofosfamide) for 6 months improves the event free survival (EFS) in patients with localised high-risk RMS and RMS-like Soft Tissue Sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent for registration, randomisation, data collection/transfer, and tumour material asservation available
* pathologically (including molecular pathology) proven diagnosis of rhabdomyosarcoma (RMS) or RMS-like soft tissue sarcoma (STS) and tumour material available for pathology review
* Rhabdomyosarcoma of the "High Risk" Group, i.e.:

  * RME, N0, M0, IRS II&III, >5 cm or >10 years in EXT, HN-PM, OTH, UG-BP
  * RME, N1, M0, any IRS-group, any size or age
  * RMA, NO, M0, any IRS-group, any size or age (exception: paratesticular RMA are not eligible) or
* Rhabdomyosarcoma of the "Very High Risk" Group, i.e.:

  * RMA, N1, MO, IRS II&III, any size or age or
  * localised high-risk RMS-like Soft Tissue Sarcoma, i.e.:
  * EES, pPNET, UDS: any N, M0, any IRS-group, any size or age
  * SySa, any N, M0, any size or age (exception: SySa IRSI&II, not T2b, N0, M0 are not eligible)
* no pre-existing illness preventing treatment (esp. those listed in the medicinal product information, e.g. cardiac, hepatic, metabolic, or renal dysfunction; hypersensitivity)
* no previous malignant tumours
* available for long term follow up through the treating centre
* in remission (according to the CWS-2007-HR definition (see X7.1.8X)) at the time of randomisation after standard multimodal therapy e.g. according to the CWS-guidance

Exclusion Criteria:

* pregnant or lactating women
* other medical condition precluding treatment with protocol therapy (e.g. HIV, psychiatric disorder, etc.)
* for sexually active females and males in Arm B (O-TIE treatment): refusal to use effective contraception (e.g. oral, IUD)

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 195 (Actual)
Dates: Start 2009-07-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
event free survival (EFS) | 3 years

SECONDARY OUTCOMES:
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Koscielniak, MD, Principal Investigator — Olgahospital, CWS; Thomas Klingebiel, MD, Study Chair — Universitätsklinikum Frankfurt, CWS; Monika Sparber Sauer, MD, Study Director — Olgahospital, CWS
Locations (87):
- Austria (8):
  - Krankenhaus der Stadt Dornbirn, Dornbirn
  - Universitätsklinik für Kinder- und Jugendheilkunde, Graz
  - Universitätsklinik für Kinder- und Jugendheilkunde, Innsbruck
  - Landeskrankenhaus, Klagenfurt
  - Landeskrankenhaus, Leoben
  - Landesfrauen - und Kinderklinik Linz, Linz
  - St. Johanns Spital / Landeskrankenhaus, Salzburg
  - St. Anna Kinderspital, Vienna
- Germany (54):
  - Universitätsklinikum, Aachen
  - Klinikum Augsburg, Augsburg
  - Charité, Berlin
  - Helios Klinikum Berlin-Buch, Berlin
  - Krankenhaus Bielefeld, Bielefeld
  - Universitätskinderklinik, Bonn
  - Klinikum Braunschweig, Braunschweig
  - Prof. Hess Kinderklinik, Bremen
  - Klinikum Chemnitz, Chemnitz
  - Kliniken der Stadt Köln, Cologne
  - Universitätsklinikum, Cologne
  - Vestische Kinderklinik, Datteln
  - Westfälisches Kinderzentrum, Klinikum Dortmund, Dortmund
  - Universitätsklinikum, Dresden
  - Universitätskinderklinik, Düsseldorf
  - Helios Klinikum, Erfurt
  - Universitätsklinikum, Erlangen
  - Universitätsklinikum, Essen
  - Universitätsklinikum, Frankfurt
  - Universitätsklinikum, Freiburg im Breisgau
  - Universitätsklinikum, Giessen
  - Universitätsklinikum, Göttingen
  - Universitätsklinikum, Greifswald
  - Universitätsklinikum, Halle
  - Universitätsklinikum, Hamburg
  - Medizinische Hochschule, Hanover
  - Universitätsklinikum, Heidelberg
  - Gemeinschaftskrankenhaus Herdecke, Herdecke
  - Universitätsklinikum, Homburg
  - Universitätsklinikum, Jena
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - Klinikum Kassel, Kassel
  - Universitätsklinikum, Kiel
  - Gemeinschaftsklinikum Mayen-Koblenz, Koblenz
  - Universitätsklinikum, Leipzig
  - Universitätsklinikum, Lübeck
  - Universitätsklinikum, Magdeburg
  - Universitätsklinikum, Mainz
  - Universitätsklinikum, Mannheim
  - Klinikum Minden, Minden
  - Dr. von Haunersches Kinderspital, München
  - Krankenhaus München Schwabing, München
  - Universitätsklinikum, Münster
  - Cnopf'sche Kinderklinik, Nuremberg
  - Klinikum Oldenburg, Oldenburg
  - Universitätsklinikum, Regensburg
  - Universitätsklinikum, Rostock
  - Asklepios Kinderklinik, Sankt Augustin
  - Helios Kliniken Schwerin, Schwerin
  - Olgahospital, Stuttgart
  - Mutterhaus der Borromäerinnen, Trier
  - Universitätsklinikum, Tübingen
  - Universitätsklinikum, Ulm
  - Universitätsklinikum, Würzburg
- Poland (10):
  - Medical University, Bialystok
  - Collegium Medicum, Bydgoszcz
  - Medical Academy, Gdansk
  - Silesian Medical Academy, Katowice
  - Polish-American Institute of Paediatrics Jagiellonian University Medical College, Krakow
  - Medical Academy, Lodz
  - Medical Academy, Lublin
  - Pian Medical University, Szczecin
  - Department of Surgical Oncology for Children and Youth, Warsaw
  - Medical University, Wroclaw
- Sweden (6):
  - Sahlgrenska University Hospital, The Queen Siliva Childrens Hospital, Gothenburg
  - University Hospital, Dept. of Pediatrics, Linköping
  - University Hospital, Dept. of Pediatric Hematology and Oncology, Lund
  - Karolinska University Hospital, Astrid Lindgrens Children's Hospital, Stockholm
  - Norrland's University Hospital, Dept. of Pediatrics, Umeå
  - Children's University Hospital, Uppsala
- Switzerland (9):
  - Kantonsspital, Aarau
  - Universitätskinderklinik beider Basel, Basel
  - Ospedale San Giovanni, Bellinzona
  - Inselspital University hospital, Bern
  - Hopital Cantonal de Geneve, Geneva
  - CHUV, Lausanne
  - Kinderspital, Lucerne
  - Ostschweizer Kinderspital, Sankt Gallen
  - University Children's Hospital, Zurich

REFERENCES:
- [Background] Dantonello TM, Int-Veen C, Harms D, Leuschner I, Schmidt BF, Herbst M, Juergens H, Scheel-Walter HG, Bielack SS, Klingebiel T, Dickerhoff R, Kirsch S, Brecht I, Schmelzle R, Greulich M, Gadner H, Greiner J, Marky I, Treuner J, Koscielniak E. Cooperative trial CWS-91 for localized soft tissue sarcoma in children, adolescents, and young adults. J Clin Oncol. 2009 Mar 20;27(9):1446-55. doi: 10.1200/JCO.2007.15.0466. Epub 2009 Feb 17. PMID 19224858
- [Background] Mattke AC, Bailey EJ, Schuck A, Dantonello T, Leuschner I, Klingebiel T, Treuner J, Koscielniak E. Does the time-point of relapse influence outcome in pediatric rhabdomyosarcomas? Pediatr Blood Cancer. 2009 Jul;52(7):772-6. doi: 10.1002/pbc.21906. PMID 19165889
- [Background] Dantonello TM, Int-Veen C, Winkler P, Leuschner I, Schuck A, Schmidt BF, Lochbuehler H, Kirsch S, Hallmen E, Veit-Friedrich I, Bielack SS, Niggli F, Kazanowska B, Ladenstein R, Wiebe T, Klingebiel T, Treuner J, Koscielniak E. Initial patient characteristics can predict pattern and risk of relapse in localized rhabdomyosarcoma. J Clin Oncol. 2008 Jan 20;26(3):406-13. doi: 10.1200/JCO.2007.12.2382. PMID 18202417
- [Background] Weihkopf T, Blettner M, Dantonello T, Jung I, Klingebiel T, Koscielniak E, Luckel M, Spix C, Kaatsch P. Incidence and time trends of soft tissue sarcomas in German children 1985-2004 - a report from the population-based German Childhood Cancer Registry. Eur J Cancer. 2008 Feb;44(3):432-40. doi: 10.1016/j.ejca.2007.11.013. PMID 18077150
- [Background] Koscielniak E, Morgan M, Treuner J. Soft tissue sarcoma in children: prognosis and management. Paediatr Drugs. 2002;4(1):21-8. doi: 10.2165/00128072-200204010-00003. PMID 11817983
- [Background] Dantonello TM, Winkler P, Boelling T, Friedel G, Schmid I, Mattke AC, Ljungman G, Bielack SS, Klingebiel T, Koscielniak E; CWS Study Group. Embryonal rhabdomyosarcoma with metastases confined to the lungs: report from the CWS Study Group. Pediatr Blood Cancer. 2011 May;56(5):725-32. doi: 10.1002/pbc.22862. Epub 2010 Nov 8. PMID 21370403
- [Background] Siepermann M, Koscielniak E, Dantonello T, Klee D, Boos J, Krefeld B, Borkhardt A, Hoehn T, Asea A, Wessalowski R. Oral low-dose chemotherapy: successful treatment of an alveolar rhabdomyosarcoma during pregnancy. Pediatr Blood Cancer. 2012 Jan;58(1):104-6. doi: 10.1002/pbc.22934. Epub 2011 Jan 16. PMID 22076833
- [Result] Klingebiel T, Boos J, Beske F, Hallmen E, Int-Veen C, Dantonello T, Treuner J, Gadner H, Marky I, Kazanowska B, Koscielniak E. Treatment of children with metastatic soft tissue sarcoma with oral maintenance compared to high dose chemotherapy: report of the HD CWS-96 trial. Pediatr Blood Cancer. 2008 Apr;50(4):739-45. doi: 10.1002/pbc.21494. PMID 18286501
- [Derived] Koscielniak E, Ljungman G, Kazanowska B, Niggli F, Sparber-Sauer M, Handgretinger R, Zimmermann M, Boos J, Blank B, Hallmen E, Teichert von Luttichau I, Schmid I, Frohlich B, Muller HL, Behnisch W, Ladenstein R, Scheer M, Vokuhl C, von Kalle T, Blattmann C, Bielack S, Klingebiel T. Maintenance therapy with trofosfamide, idarubicin and etoposide in patients with rhabdomyosarcoma and other high-risk soft tissue sarcomas (CWS-2007-HR): a multicentre, open-label, randomised controlled phase 3 trial. EClinicalMedicine. 2024 Nov 29;78:102957. doi: 10.1016/j.eclinm.2024.102957. eCollection 2024 Dec. PMID 39687431
- See also: Related Info — http://www.kinderkrebsinfo.de/
- See also: homepage of CWS Study Group — http://cws.olgahospital-stuttgart.de